CLINICAL TRIAL: NCT05745610
Title: An Clinical Trial on the Efficacy and Safety of Shen Hai Long Capsule in the Treatment of Male Asthenospermia
Brief Title: Shen Hai Long Capsule for Male Asthenospermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yuanzhen Zhang, Prof, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shenhailong2023
Record Dates: First submitted 2023-02-13; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Efficacy and Safety of Shen Hai Long Capsule for Mild to Moderate Asthenospermia in Men
Keywords: efficacy; safety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shen Hai Long Group (Experimental)
  Interventions: Drug: Shen Hai Long Capsule
- Sheng Jing Group (Active Comparator)
  Interventions: Drug: Sheng Jing Capsule

INTERVENTIONS:
Drug: Shen Hai Long Capsule — 3 times/day (9 capsules/day) for 12 weeks
  Arms: Shen Hai Long Group
Drug: Sheng Jing Capsule — 3 times/day (12 capsules/day) for 12 weeks
  Arms: Sheng Jing Group

SUMMARY:
To evaluate the efficacy and safety of Shen Hai Long Capsule in the treatment of mild to moderate asthenospermia in men.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of Shen Hai Long Capsule in the treatment of mild to moderate asthenospermia in men: 1) Efficacy index (1) Main efficacy indexes Forward motile sperm ratio (PR) (2) Secondary efficacy indexes 1. Sperm survival rate; 2. Sperm concentration; 3. Normal morphology rate of sperm; 4. Seminal malondialdehyde (MDA) 5. Seminal superoxide dismutase (SOD) 2) Safety indicators

(1) Vital signs; (2) liver and kidney function; (3) blood routine; (4) electrocardiogram; (5) Adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 22 to 50 years old;
2. Patients with mild to moderate asthenospermia, that is, at least two normative semen analyses indicated that 10%≤PR percentage < 32% and the total number of PR sperm ranged from 5 million to 20 million;
3. At least two standard semen analyses indicated that sperm concentration ≥15×106 /ml; Sperm normal morphology rate ≥4%;
4. No other Chinese and Western drugs for the treatment of oligospermia, weak and malformed spermia have been taken in the past 3 months;
5. The subject voluntarily participates and signs the informed consent.

Exclusion Criteria:

1. Varicocele, ejaculatory duct/seminal vesicle cyst, anti-sperm antibody (+);
2. Genital tract infection: seminal plasmic elastase > 1000ng/ml or leukocyte semen disease (peroxidase positive cell concentration in semen more than 1×10^6/mL);
3. Erectile dysfunction, ejaculation disorders;
4. suffer from mental disorders, immune system diseases; Severe impairment of liver and kidney function (serum transaminase ≥2× upper limit of medical reference value, creatinine clearance ≤40ml/min or active stage of chronic kidney disease);
5. Patients with allergic history or constitution to therapeutic drugs;
6. Patients who have taken drugs affecting the study within 3 months, such as antitumor and antiepileptic drugs, etc.

Ages: 22 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Forward motile sperm ratio (PR) | 12 weeks
  To compare the PR between baseline and 12 weeks

SECONDARY OUTCOMES:
Sperm survival rate | 12 weeks
  To compare the Sperm survival rate between baseline and 12 weeks
Sperm concentration | 12 weeks
  To compare the Sperm concentration between baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuanzhen Zhang, Prof., Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Please contact the Central Contact Person for detailed study data.